CLINICAL TRIAL: NCT05894785
Title: External Cephalic Version (ECV) for Twins With Non-vertex Presenting Twin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Zvi Ehrlich, Principal Investigator, Shaare Zedek Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0327-21-SZMC
Record Dates: First submitted 2023-05-29; First posted 2023-06-08 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Twin Pregnancy With Antenatal Problem
MeSH Terms: interventions — Version, Fetal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental)
  Interventions: Procedure: External cephalic version

INTERVENTIONS:
Procedure: External cephalic version — An ECV attempt is made on the study group

SUMMARY:
In this study, women with a twin pregnancy with the presenting twin in a non-vertex(head) presenting twin undergo an external cephalic version.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older multiparous no previous cesarean delivery (CD) a non-vertex presenting twin in a term (37 weeks gestation and onwards) dichorionic diamniotic twin pregnancy

Exclusion Criteria:

* contraindication for a vaginal delivery nulliparous monochorionic diamniotic pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-27 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Success rates of ECV | 1 day

SECONDARY OUTCOMES:
Maternal and fetal morbidities | up to 7 days from enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided